CLINICAL TRIAL: NCT05006378
Title: Effect of Chamomile Intake on Blood Coagulation Tests in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Jonathon Schwartz, Clinical Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: IRB2021-00314
Record Dates: First submitted 2021-07-27; First posted 2021-08-16 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Coagulation Disorder
Keywords: Coagulation; Chamomile
MeSH Terms: conditions — Hemostatic Disorders; Thrombosis | interventions — Chamomile extract

STUDY DESIGN:
Intervention Model Description: This is a placebo-controlled complete crossover study with 3 treatments: (A) placebo, (B) chamomile extract capsule, and (C) chamomile tea. Every participant will receive all three treatments. There are 6 possible sequences of treatment (ABC, ACB, BAC, BCA, CAB, CBA). Blocked randomization lists for sequence assignment will be computed using statistical software. Each participant will be randomly assigned one of the six treatment sequences using REDCap software. Carryover effects will be minimized by maintaining a consistent washout time of 1 week between treatments. Blood sampling will be conducted immediately before and after the treatment weeks.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo Capsule (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Capsule
- Chamomile Tea (Experimental): Subjects will consume three servings of chamomile tea throughout the day for the one-week treatment period. Each tea serving will be prepared using 3 grams of chamomile tea steeped in hot water according to the study protocol.
  Interventions: Dietary Supplement: Chamomile Tea
- Chamomile Extract Capsule (Experimental): Subjects will consume three chamomile capsules throughout the day for the one-week treatment period. Each capsule consists of 500 milligrams of a chamomile extract that has been standardized to 1.2% apigenin content.
  Interventions: Dietary Supplement: Chamomile Extract Capsule

INTERVENTIONS:
Dietary Supplement: Chamomile Tea — Chamomile tea bags consumed by subjects as described in study arms section.
  Arms: Chamomile Tea
Dietary Supplement: Chamomile Extract Capsule — Chamomile extract capsules consumed by subjects as described in "Experimental: Chamomile Extract Capsule" study arms section.
  Arms: Chamomile Extract Capsule
Dietary Supplement: Placebo Capsule — Placebo capsules consumed by subjects as described in "Placebo Comparator" study arms section.
  Arms: Placebo Capsule

SUMMARY:
Chamomile may possess anticoagulant effects based on the presence of coumarin-like compounds within the flower. This randomized, placebo-controlled complete crossover study will investigate the impact of chamomile ingestion on coagulation.

DETAILED DESCRIPTION:
Subjects will be enrolled into three groups in a crossover fashion upon obtaining written informed consent. Baseline laboratory screening assays of anticoagulation will be obtained. The three intervention groups include (1) chamomile tea intake, (2) chamomile extract intake and (3) placebo capsules. Subjects will consume the chamomile or placebo preparations for one week and partake in a one-week washout period between interventions. Screening assays of coagulation will be obtained immediately before and after each intervention week.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed written consent
* Able to withhold use of other chamomile products (teas, lotions, supplements, extracts); will only use study-supplied chamomile products.

Exclusion Criteria:

* Past medical/family history of bleeding/thrombotic disorders (e.g. hemophilia, von-Willebrand disease)
* Chronic medications known to affect hemostasis (anticoagulants, antiplatelet agents, SSRIs, herbal/complementary medicine agents)
* Three or more alcoholic drinks daily
* Sedentary status/ restricted mobility
* Active smoker or quit smoking within one week of screening
* Females who are pregnant, breast-feeding, or lactating
* Scheduled surgical procedure during study period
* Hospitalized patients
* Underweight (BMI < 18 kg/m2) or history of malnourishment
* Active symptoms of a respiratory, dermatologic, urinary, or gastrointestinal infection
* Diagnosed allergy to chamomile
* Severe allergy to ragweed
* Physical inability to consume chamomile tea according to the study dosing schedule
* Prescription usage of an anticoagulant agent such as warfarin, anti-Xa inhibitor, or other novel oral anticoagulants
* ADP antagonist use, including clopidogrel, prasugrel, and ticagrelor
* GPIIb/IIIa inhibitor use, including ticlopidine, eptifibatide
* More than weekly NSAID use (e.g. aspirin, ibuprofen, naproxen)
* Diagnosis of a bleeding-diathesis disorder
* Diagnosis of a hypercoagulable state
* History of elevated INR (including baseline study) or other abnormal bleeding study (PT, aPTT, thrombin time, reptilase time, above the upper limit of normal for Stony Brook Hospital Reference Range) while not taking anticoagulants or herbal supplements listed below
* Active intake of the following herbal supplements at time of study enrollment that may alter baseline coagulation function including:

  * Ginger
  * Garlic
  * Gingko
  * Ginseng
  * Fish oil
  * Black Cohosh
  * Feverfew
  * Valerian
  * Coenzyme Q10
  * Goldenseal
  * St. John Wort
* Baseline CBC with either a hematocrit below 30% or platelet count below 150,000, white blood cell count above 15,000 or less than 3,000.
* Inability to discontinue the aforementioned herbal supplements more than 14 days before enrollment into the study.
* History of estrogen-dependent condition such as uterine fibroids, breast cancer, uterine cancer, or ovarian cancer
* Significant fear of needles or fainting blood draws
* Actively taking cyclosporine
* Patient refusal to participate in study for the allotted study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Change in Prothrombin Time | One week following each treatment

SECONDARY OUTCOMES:
Change in Activated Partial Thromboplastin Time | One week following each treatment
Change in Thrombin Time | One week following each treatment
Change in Reptilase Time | One week following each treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwartz JA, Romeiser JL, Kimura R, Senzel L, Galanakis D, Halper D, Mena S, Bennett-Guerrero E. Effect of chamomile intake on blood coagulation tests in healthy volunteers: a randomized, placebo-controlled, crossover trial. Perioper Med (Lond). 2023 Sep 20;12(1):51. doi: 10.1186/s13741-023-00339-7. PMID 37730613